CLINICAL TRIAL: NCT05353491
Title: Technology-assisted Cognitive-behaviour Therapy Delivered by Peers Versus Standard Cognitive Behaviour Therapy Delivered by Community Health Workers for Perinatal Depression: A Cluster Randomised Controlled Non-inferiority Trial
Brief Title: Thinking Healthy Program-Technology Assisted (THP-TA)
Acronym: THP-TA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: Shifa Tameer-e-Millat University (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Siham Sikander, Co-investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UoL001668; NIHR200817 (Other Grant/Funding Number: National Institute for Health Research, UK)
Record Dates: First submitted 2022-03-28; First posted 2022-04-29 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Perinatal Depression; Depression, Postpartum
Keywords: Perinatal depression; Perinatal anxiety; perinatal mental health conditions; electronic CBT; CBT; task shifting; low-resourced settings; task sharing; Thinking Healthy Programme; LMIC; Technology-assisted; peers; community health workers
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology assisted Thinking Healthy Program delivered by peers (Experimental): A technology adapted version of the Thinking Healthy Program (THP) delivered by peers using multimedia android based app. The bespoke android app leverages human-centered design and makes use of 2-d videos demonstrating narrative scripts delivered by culturally appropriate animated avatars representing depressed mothers, families, peers and mental health experts.
  It is designed as a low intensity psychosocial multicomponent intervention based on cognitive behavioral approaches. The THP improves depression through psychoeducation, behavior activation, thought challenging, improving problem solving skills and by activating social support networks.
  The intervention program comprises of 8 sessions delivered by trained peers.
  Interventions: Behavioral: Technology assisted Thinking Healthy Program (THP-TA)
- Standard Thinking Healthy Program delivered by community health workers (Active Comparator): The Thinking Healthy Programme (THP) is a CBT-based manualised paper version of the intervention targeting women with perinatal depression in low socioeconomic settings.
  The CBT techniques include guided discovery using illustrated brief vignettes, behavioural activation, and problem solving. Non-specific techniques include empathic listening and promoting social support from key family members for the mother in negotiating challenges during the perinatal period. This intervention programme is paper based utilizing reference manual, health calendar and job aid as tools for delivering content.
  The intervention employs these techniques to improve outcomes in three areas: maternal well-being, mother-infant interaction and relationship with significant others. The intervention consists of 8 core sessions starting in the second or third trimester of pregnancy and continuing to 3 months postnatal.
  Interventions: Behavioral: Standard Thinking Healthy Program

INTERVENTIONS:
Behavioral: Technology assisted Thinking Healthy Program (THP-TA) — A technology adapted version of the Thinking Healthy Program (THP) delivered by peers using multimedia android based app.
  Arms: Technology assisted Thinking Healthy Program delivered by peers
Behavioral: Standard Thinking Healthy Program — This intervention paper-based manual delivered by lady health workers ie government employed community health workers with health training background.
  Arms: Standard Thinking Healthy Program delivered by community health workers

SUMMARY:
Background

The Thinking Healthy Program (THP) is an evidence based task-shifted low intensity psychosocial intervention, recommended by the World Health Organization for the treatment of perinatal depression. The investigators developed a technology-assisted version of Thinking Healthy Program (THP-TA) which allows peers to deliver the THP, while ensuring minimal resources for training of delivery agents and ensuring adequate fidelity.

Method

This is a non-inferiority, pragmatic cluster randomized controlled trial designed to test the primary hypothesis that technology assisted delivery of THP is not worse than THP intervention delivered by community health workers, in increasing perinatal depression remission rates at 3 months postnatal. In addition, this study will also test the effectiveness of the THP-TA in improving recovery from perinatal depression at 6 months postpartum, quality of life and social support. This study also aims to evaluate the cost-effectiveness of the THP-TA.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with current major depressive episode in their second or third trimester (4 to 8 months of pregnancy).
2. Aged 18 years and above
3. Intent to stay in the study area for at least 1 year.

Exclusion Criteria:

1. Women requiring inpatient care for any reason (medical or psychiatric) as determined by their primary health care professional
2. Those who do not comprehend Urdu language will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 980 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Remission rates of perinatal depression | 3 months postnatal
  Remission rates from perinatal depression among the trial participants will be based on clinical diagnostic criteria based on the Structured Clinical Interview for the DSM-IV Axis (SCID) module. The SCID will be employed at baseline and 3 months postnatal.

SECONDARY OUTCOMES:
Sustained remission rates of perinatal depression | 3 months and 6 months postnatal
  Sustained remission rates from perinatal depression among the trial participants will be based on clinical diagnostic criteria based on the Structured Clinical Interview for the DSM-IV Axis (SCID) module, assessed at baseline, 3 and 6 months postnatal.
Change in severity of perinatal depressive symptoms | 3 months and 6 months postnatal
  Severity of perinatal depressive symptoms will be measured using the Patient Health Questionnaire-9 items assessed at baseline, 3 months and 6 months postnatal. Score on this scale ranges from 0 to 27, with higher scores indicating increased severity.
Change in severity of perinatal anxiety symptoms | 3 months and 6 months postnatal
  Severity of perinatal anxiety symptoms will be measured using the Generalized anxiety Disorder-7 scale assessed at baseline, 3 months and 6 months postnatal. Score on this scale ranges from 0 to 21, with higher scores indicating increased severity.
Change in maternal Quality of Life | 3 months and 6 months postnatal
  Change in maternal quality of life will be measured using the EuroQuality of Life scale (EQ-5D-3L), at baseline, 3 months and 6 months postnatal. It is a valid and reliable scale to quantify health status across 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change in disability using the World Health Organization Disability Assessment Schedule 2.0 | 3 months and 6 months postnatal
  This World Health Organization Disability Assessment Schedule 2.0 questionnaire assesses disability due to health conditions or illnesses (chronic or acute) including mental and emotional health problems. It is a valid and reliable instrument that generates domain-specific scores for six different functioning domains: i) cognition ii) mobility iii) self-care iv) getting along v) life activities (household and work/school) and vi) participation. It will be employed at baseline, 3 and 6 months postnatal.
Service use and costs | Pregnancy through to 6 months postnatal
  Service use will be measured using Client Service Receipt Inventory (CSRI), including costs of healthcare services used, details and costs of medications and wider health service utilization and economic costs at 3 months and 6 months postnatal.
Infant nutrition/breastfeeding | 3 months and 6 months postnatal
  Using 24-hour recall WHO breastfeeding practices tool, we will quantify percentage of infants being exclusively breastfed at 3 months and 6 months postnatal.
Family planning practices | 3 months and 6 months postnatal
  To ascertain family planning practices, categorical questions will be asked regarding the use of contraception during the postpartum period.
Infant Immunization Status | 3 months and 6 months postnatal
  Immunization status of the infant will be assessed using a categorical question assessing completely or incompletely immunized as per the Expanded Programme on Immunization program in Pakistan, at 3 months and 6 months postnatal.
Maternal Social support | 3 months and 6 months postnatal
  Multidimensional Scale of Perceived Social Support (MSPSS) will be used to assess the perceived levels of social support among the intervention recipients at baseline, 3 months and 6 months postnatal, from three sources: family, friends and significant other. It comprises of 12 items, scores on which can be summed together with higher scores corresponding to better social support.
Parental time spent in play with the infant | 3 months and 6 months postnatal
  Parental time spent in play with the infant will be assessed at 3 months and 6 months postnatal.
Diarrheal episodes among infants | 3 months and 6 months postnatal
  Number of episodes of diarrheal episodes among infants will be assessed using the WHO criteria and definitions, at 3 months and 6 months postnatal
Acute upper respiratory tract infections among infants | 3 months and 6 months postnatal
  Number of episodes of acute upper respiratory tract infections among infants will be assessed using the WHO criteria and definitions, at 3 months and 6 months postnatal

CONTACTS AND LOCATIONS:
Locations (1):
- Human Development Research Foundation, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
After the publication of results focusing on primary and secondary outcomes/endpoints, anonymous data can be made available to researchers who provide a methodologically sound proposal, on request.

REFERENCES:
- [Background] Rahman A, Malik A, Sikander S, Roberts C, Creed F. Cognitive behaviour therapy-based intervention by community health workers for mothers with depression and their infants in rural Pakistan: a cluster-randomised controlled trial. Lancet. 2008 Sep 13;372(9642):902-9. doi: 10.1016/S0140-6736(08)61400-2. PMID 18790313
- [Background] Sikander S, Ahmad I, Atif N, Zaidi A, Vanobberghen F, Weiss HA, Nisar A, Tabana H, Ain QU, Bibi A, Bilal S, Bibi T, Liaqat R, Sharif M, Zulfiqar S, Fuhr DC, Price LN, Patel V, Rahman A. Delivering the Thinking Healthy Programme for perinatal depression through volunteer peers: a cluster randomised controlled trial in Pakistan. Lancet Psychiatry. 2019 Feb;6(2):128-139. doi: 10.1016/S2215-0366(18)30467-X. PMID 30686386
- [Background] Fuhr DC, Weobong B, Lazarus A, Vanobberghen F, Weiss HA, Singla DR, Tabana H, Afonso E, De Sa A, D'Souza E, Joshi A, Korgaonkar P, Krishna R, Price LN, Rahman A, Patel V. Delivering the Thinking Healthy Programme for perinatal depression through peers: an individually randomised controlled trial in India. Lancet Psychiatry. 2019 Feb;6(2):115-127. doi: 10.1016/S2215-0366(18)30466-8. PMID 30686385
- [Background] Rahman A, Akhtar P, Hamdani SU, Atif N, Nazir H, Uddin I, Nisar A, Huma Z, Maselko J, Sikander S, Zafar S. Using technology to scale-up training and supervision of community health workers in the psychosocial management of perinatal depression: a non-inferiority, randomized controlled trial. Glob Ment Health (Camb). 2019 May 16;6:e8. doi: 10.1017/gmh.2019.7. eCollection 2019. PMID 31157115
- [Background] Maselko J, Sikander S, Turner EL, Bates LM, Ahmad I, Atif N, Baranov V, Bhalotra S, Bibi A, Bibi T, Bilal S, Biroli P, Chung E, Gallis JA, Hagaman A, Jamil A, LeMasters K, O'Donnell K, Scherer E, Sharif M, Waqas A, Zaidi A, Zulfiqar S, Rahman A. Effectiveness of a peer-delivered, psychosocial intervention on maternal depression and child development at 3 years postnatal: a cluster randomised trial in Pakistan. Lancet Psychiatry. 2020 Sep;7(9):775-787. doi: 10.1016/S2215-0366(20)30258-3. PMID 32828167
- [Background] Vanobberghen F, Weiss HA, Fuhr DC, Sikander S, Afonso E, Ahmad I, Atif N, Bibi A, Bibi T, Bilal S, De Sa A, D'Souza E, Joshi A, Korgaonkar P, Krishna R, Lazarus A, Liaqat R, Sharif M, Weobong B, Zaidi A, Zuliqar S, Patel V, Rahman A. Effectiveness of the Thinking Healthy Programme for perinatal depression delivered through peers: Pooled analysis of two randomized controlled trials in India and Pakistan. J Affect Disord. 2020 Mar 15;265:660-668. doi: 10.1016/j.jad.2019.11.110. Epub 2019 Nov 23. PMID 32090783
- [Derived] Rahman A, Malik A, Nazir H, Zaidi A, Nisar A, Waqas A, Atif N, Gibbs NK, Luo Y, Sikander S, Wang D. Technology-assisted cognitive-behavioral therapy for perinatal depression delivered by lived-experience peers: a cluster-randomized noninferiority trial. Nat Med. 2025 Jul;31(7):2196-2203. doi: 10.1038/s41591-025-03655-1. Epub 2025 Apr 8. PMID 40200057
- [Derived] Rahman A, Malik A, Atif N, Nazir H, Zaidi A, Nisar A, Waqas A, Sharif M, Chen T, Wang D, Sikander S. Technology-assisted cognitive-behavior therapy delivered by peers versus standard cognitive behavior therapy delivered by community health workers for perinatal depression: study protocol of a cluster randomized controlled non-inferiority trial. Trials. 2023 Aug 25;24(1):555. doi: 10.1186/s13063-023-07581-w. PMID 37626428

DOCUMENTS (1):
  • Informed Consent Form (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT05353491/ICF_000.pdf